CLINICAL TRIAL: NCT00529217
Title: Treatment of Depersonalization Disorder With Transcranial Magnetic Stimulation (TMS)
Acronym: TMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5269
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2013-11

CONDITIONS: Depersonalization Disorder
Keywords: Dissociative; Dissociation; Depersonalization; Depersonalization Disorder; Transcranial Magnetic Stimulation; TMS; Depersonalization Disorder (DPD); rTMS
MeSH Terms: conditions — Depersonalization; Dissociative Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-Label Active rTMS (Experimental): Active repetitive Transcranial Magnetic Stimulation (rTMS)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Strong electromagnetic fields (~2Tesla) generated briefly (~1ms) but repetitively (1Hz) applied for 30mins, in five sessions per week for up to twelve weeks.
  Other Names: Magstim, Magstim Rapid, Magstim Rapid2

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of transcranial magnetic stimulation in the treatment of Depersonalization Disorder (DPD).

DETAILED DESCRIPTION:
This study is a research trial of an outpatient, non-medication, non-invasive investigational treatment called Transcranial Magnetic Stimulation (TMS). TMS applies a magnetic field to the brain for a brief period of time. TMS is a procedure that involves 30 minute-long daily sessions every weekday for a series of weeks. The investigators are testing whether TMS can treat Depersonalization Disorder (DPD).

This is an open-label study. All patients will receive active treatment. DPD symptoms will be monitored through weekly self-report questionnaires as well clinical ratings with a doctor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients, 18 to 70 years of age.
* Primary diagnosis of Depersonalization Disorder.
* Duration of the index episode of at least a year.
* Patients currently on DPD medication must be at the same stable dose(s) at least 2 months and be to continue at the same dose(s) through the duration of the study.
* Capable and willing to provide informed consent

Exclusion Criteria:

* Individuals with a neurological disorder including, but not limited to: brain lesion; history of seizures; history of cerebrovascular accident; history of stroke; cerebral aneurysm, Dementia; Parkinson's Disease; Huntington's chorea; Multiple Sclerosis.
* Increased risk of seizure for any reason, including prior head trauma with loss of consciousness for 5 minutes or more.
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease.
* Intracranial implants (e.g. aneurysms clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
* If participating in psychotherapy, must have been in stable treatment for at least three months prior to entry into the study, with no anticipation of change in frequency of therapeutic sessions, or the therapeutic focus over the duration of the rTMS trial.
* Known or suspected pregnancy.
* Women who are breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-05; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Mantovani, MD, Principal Investigator — Columbia
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Blanke O, Mohr C, Michel CM, Pascual-Leone A, Brugger P, Seeck M, Landis T, Thut G. Linking out-of-body experience and self processing to mental own-body imagery at the temporoparietal junction. J Neurosci. 2005 Jan 19;25(3):550-7. doi: 10.1523/JNEUROSCI.2612-04.2005. PMID 15659590
- [Background] Chen R, Classen J, Gerloff C, Celnik P, Wassermann EM, Hallett M, Cohen LG. Depression of motor cortex excitability by low-frequency transcranial magnetic stimulation. Neurology. 1997 May;48(5):1398-403. doi: 10.1212/wnl.48.5.1398. PMID 9153480
- [Background] Hunter EC, Baker D, Phillips ML, Sierra M, David AS. Cognitive-behaviour therapy for depersonalisation disorder: an open study. Behav Res Ther. 2005 Sep;43(9):1121-30. doi: 10.1016/j.brat.2004.08.003. PMID 16005701
- [Background] Jimenez-Genchi AM. Repetitive transcranial magnetic stimulation improves depersonalization: a case report. CNS Spectr. 2004 May;9(5):375-6. doi: 10.1017/s1092852900009366. PMID 15115950
- [Background] Sierra M, Phillips ML, Ivin G, Krystal J, David AS. A placebo-controlled, cross-over trial of lamotrigine in depersonalization disorder. J Psychopharmacol. 2003 Mar;17(1):103-5. doi: 10.1177/0269881103017001712. PMID 12680746
- [Background] Simeon D, Guralnik O, Hazlett EA, Spiegel-Cohen J, Hollander E, Buchsbaum MS. Feeling unreal: a PET study of depersonalization disorder. Am J Psychiatry. 2000 Nov;157(11):1782-8. doi: 10.1176/appi.ajp.157.11.1782. PMID 11058475
- [Background] Simeon D, Guralnik O, Schmeidler J, Knutelska M. Fluoxetine therapy in depersonalisation disorder: randomised controlled trial. Br J Psychiatry. 2004 Jul;185:31-6. doi: 10.1192/bjp.185.1.31. PMID 15231553
- [Background] Simeon D, Knutelska M. An open trial of naltrexone in the treatment of depersonalization disorder. J Clin Psychopharmacol. 2005 Jun;25(3):267-70. doi: 10.1097/01.jcp.0000162803.61700.4f. PMID 15876908
- [Background] Simeon D. Depersonalisation disorder: a contemporary overview. CNS Drugs. 2004;18(6):343-54. doi: 10.2165/00023210-200418060-00002. PMID 15089102
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- See also: Division of Brain Stimulation and Therapeutic Modulation web site — http://www.brainstimulation.columbia.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Brain Behavior Clinic of Columbia Psychiatry and the Depersonalization and Dissociation Program of Mount Sinai and Beth Israel Medical Centers in New York.
Pre-assignment Details: No enrolled participant was excluded from the trial. Twelve outpatients entered the study.
Groups:
- Open-Label, rTMS, Active Coil: Repetitive Transcranial Magnetic Stimulation (rTMS) : Strong electromagnetic fields (~2Tesla) generated briefly (~1ms) but repetitively (1Hz) applied for 30mins, in five sessions per week for up to twelve weeks.
Period: Overall Study
Arm/Group | Open-Label, rTMS, Active Coil
Started | 12
Completed | 8
Not Completed | 4
Not completed — Lack of Efficacy | 2
Not completed — Unable to adhere to study schedule | 2

BASELINE CHARACTERISTICS:
Groups:
- Open-Label Active: Repetitive Transcranial Magnetic Stimulation (rTMS) : Strong electromagnetic fields (~2Tesla) generated briefly (~1ms) but repetitively (1Hz) applied for 30mins, in five sessions per week for up to twelve weeks.
Arm/Group | Open-Label Active
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Cambridge Depersonalization Scale (CDS)
Description: Change on CDS from baseline. Scale item number: 29 Item score range: Frequency: 0 - 4, Duration: 0-5 Minimum CDS score: 0 Maximum CDS score: 261
  Higher scores indicate the presence of high symptom severity. Decrease in scores from baseline reflects clinical symptom improvement.
Time Frame: 6, 9, or 12 weeks
Measure: Number; unit: responders (>50% reduction in CDS score)
Arm/Group | Open-Label, rTMS, Active Coil
Number analyzed (Participants) | 12
responders (>50% reduction in CDS score) | 6

2. Secondary Outcome: Clinical Improvement (CGI-S)
Description: Minimum CGI-S score: 1 Maximum CGI-S score: 7
  Higher scores indicate the presence of high symptom severity. Decrease in scores from baseline reflects clinical symptom improvement.
  Patients will be classified as responders with a CGI-S = 1 or 2; and partial responders CGI-S = 3.
  1. = Normal, not at all ill
  2. = Borderline mentally ill
  3. = Mildly ill
  4. = Moderately ill
  5. = Markedly ill
  6. = Severely ill
  7. = Among the most extremely ill patients
Time Frame: 6, 9, or 12 weeks
Measure: Number; unit: responders (CGI-S = 1 or 2)
Arm/Group | Open-Label Active
Number analyzed (Participants) | 12
responders (CGI-S = 1 or 2) | 6

ADVERSE EVENTS:
Arm/Group | Open-Label Active
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes